CLINICAL TRIAL: NCT06836089
Title: DWI Breast MRI in Dense Breast: A Clinical Trial to Assess the Efficacy and Diagnostic Accuracy of Diffusion Weighted Imaging in Dense Breast Tissue
Acronym: DWI-Breast MRI
Status: Enrolling by invitation | Type: Observational
Sponsor: Graziella di Grezia (Other)
Collaborators: Link Campus University (Other); University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor-Investigator, Graziella di Grezia, Principal Investigator, Link Campus University
Organization: Link Campus University (Other)
Other Study IDs: T_3_2025
Record Dates: First submitted 2025-02-15; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Dense Breast Parenchyma; Breast Cancer Detection; DWI
Keywords: Breast MRI; DWI; dense breast

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group of women with dense breast

SUMMARY:
his clinical trial aims to evaluate the efficacy and diagnostic accuracy of Diffusion Weighted Imaging (DWI) in breast MRI for women with dense breast tissue. DWI is investigated as an adjunctive method to improve early tumor detection in women with dense breasts, a group at high risk for delayed diagnosis due to limited visibility in mammography.

Study Purpose:

To assess the utility of Diffusion Weighted Imaging (DWI) in improving diagnostic accuracy for patients with dense breasts.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 40-75 years.
* Patients with dense breast tissue, classified according to BI-RADS (Breast Imaging-Reporting and Data System).
* Patients who previously underwent breast MRI, including Diffusion Weighted Imaging (DWI).
* Availability of histopathological confirmation for breast lesions (biopsy results).

Exclusion Criteria:

* Patients with a known allergy to gadolinium-based contrast agents.
* Pregnant or breastfeeding women at the time of imaging.
* Presence of metallic implants or other MRI-incompatible devices.
* Patients with incomplete imaging datasets (e.g., missing DWI sequences or non-standardized protocols).
* Prior history of breast cancer treatment (surgery, chemotherapy, or radiotherapy) before the imaging study.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will analyze a retrospective cohort of women aged 40-75 years with dense breast tissue, classified according to BI-RADS criteria. The population consists of patients who previously underwent breast MRI with Diffusion Weighted Imaging (DWI) as part of their clinical evaluation for breast cancer screening or diagnostic workup.
  The dataset includes cases from multiple imaging centers, ensuring variability in patient demographics and imaging protocols. The study population will encompass:
  Women with dense breasts, a group at higher risk for missed diagnoses due to the limitations of mammography.
  Patients with both benign and malignant breast lesions, confirmed through histopathology (biopsy results).
  Cases where mammography, tomosynthesis, and conventional MRI were performed, allowing for a comparative diagnostic accuracy assessment.
  Patients with prior breast cancer treatment, missing imaging sequences, or MRI-incompatible conditions will be excluded to maintain data consiste
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Diffusion Weighted Imaging (DWI) in Dense Breast Tissue: A Retrospective Cohort Study | 12 months
  This retrospective cohort study aims to assess the diagnostic accuracy and clinical utility of Diffusion Weighted Imaging (DWI) in breast MRI for women with dense breast tissue. By analyzing previously collected imaging data, the study evaluates the sensitivity, specificity, and predictive value of DWI in detecting malignant breast lesions. The research also examines the correlation between Apparent Diffusion Coefficient (ADC) values and histopathological tumor characteristics, comparing DWI's performance with conventional MRI and mammography/tomosynthesis.

CONTACTS AND LOCATIONS:
Overall Officials: Graziella Di Grezia, medicine and surgery, Principal Investigator — Link Campus University; Gianluca Gatta, medicine and surgery, Study Chair — University of Campania Luigi Vanvitelli
Locations (1):
- University of Campania Luigi Vanvitelli, Naples, Italy

IPD SHARING:
Plan to Share IPD: No